CLINICAL TRIAL: NCT03188939
Title: Randomized Comparative Study Between Single-injection , Intra- Cluster -Injection and Double-injection Ultrasound-guided Supraclavicular Block of Brachial Plexus
Brief Title: Comparative Study Between Single , Intra- Cluster and Double-injection Ultrasound-guided Supraclavicular Block of Brachial Plexus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Refaat, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-34-2017
Record Dates: First submitted 2017-06-10; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Intervention Model Description: For the 3 techniques , we will prepare 20 gauge 10cm block needle and portable ultrasound machine , In single-injection technique using in plane method and lateral to medial direction, local anesthetic is injected at the point where the subclavian artery meets the first rib. In intra- cluster-injection technique using in plane method and lateral to medial direction , the local anesthetic is injected inside main and satellite neural cluster.
  In double-injection technique using in plane method and lateral to medial direction half the volume of local anesthetic is injected at intersection of first rib and subclavian artery and another half is injected supero- lateral to subclavian artery to assure spread of the local anesthetic solution in all planes containing brachial plexus.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G s (Active Comparator): 20 guage 10cm block needle inserted in the supraclavicular fossa guided by portable ultrasound machine using in plane method and lateral to medial direction, local anesthetic (30 ml bupivacaine) is injected at the point where the subclavian artery meets the first rib
  Interventions: Procedure: single injection supraclavicular brachial pleuxus block
- G ic (Active Comparator): 20 guage 10cm block needle inserted in the supraclavicular fossa guided by portable ultrasound machine using in plane method and lateral to medial direction,the local anesthetic(30 ml bupivacaine) is injected inside main and satellite neural cluster.( Circumferential administration of local anesthetic rather than creating a single point injection )
  Interventions: Procedure: intracluster injection supraclavicular brachial pieuxus block
- G d (Active Comparator): 20 guage 10cm block needle inserted in the supraclavicular fossa guided by portable ultrasound machine using in plane method and lateral to medial direction,half the volume of local anesthetic(15 ml bupivacaine) is injected at intersection of first rib and subclavian artery and another half(15 ml bupivacaine) is injected supero- lateral to subclavian artery to assure spread of the local anesthetic solution in all planes containing brachial plexus
  Interventions: Procedure: double injection supraclavicular brachial pleuxus block

INTERVENTIONS:
Procedure: single injection supraclavicular brachial pleuxus block — the investigator will prepare 20 gauge 10cm block needle and portable ultrasound machine , In single-injection technique using in plane method and lateral to medial direction, local anesthetic is injected at the point where the subclavian artery meets the first rib.
  Arms: G s
Procedure: intracluster injection supraclavicular brachial pieuxus block — the investigator will prepare 20 gauge 10cm block needle and portable ultrasound machine (Siemens ACUSON X300 Ultrasound System with linear probe 8-14 MHZ).using in plane method and lateral to medial direction , the local anesthetic(30 ml bupivacaine) is injected inside main and satellite neural cluster.( Circumferential administration of local anesthetic rather than creating a single point injection )
  Arms: G ic
Procedure: double injection supraclavicular brachial pleuxus block — the investigator will prepare 20 gauge 10cm block needle and portable ultrasound machine (Siemens ACUSON X300 Ultrasound System with linear probe 8-14 MHZ).using in plane method and lateral to medial direction , half the volume of local anesthetic(15 ml bupivacaine) is injected at intersection of first rib and subclavian artery and another half(15 ml bupivacaine) is injected supero- lateral to subclavian artery to assure spread of the local anesthetic solution in all planes containing brachial plexus
  Arms: G d

SUMMARY:
Supraclavicular block of brachial plexus is a type of regional anesthesia sometimes employed as an alternative to general anesthesia for surgery of the forearm. Many approaches have been described for ultrasound-guided supraclavicular block of the brachial plexus , Double- injection technique , single-injection and intra- cluster-injection technique. In intra- cluster-injection technique.The comparison between the 3 techniques may allow detecting the most beneficial one. the investigators hypothesized that intra-cluster-injection technique will be associated with more rapid onset, longer duration and the least complications. (because the trunks and divisions of the brachial plexus are relatively close as they travel over the first rib, the onset and quality of anesthesia will be faster and complete) Methods : This study will be conducted at kasr al ainy Hospital Cairo university After obtaining ethics committee approval and written informed consent 36 patients (who will undergo surgery for forearm)included in the study classified into three groups Gs single injection technique ,Gic intra- cluster injection technique, Gd double injection technique After block will be done, a second investigator will examine the patient for sensory and motor block (every 10 minutes for 30 minutes) and for occurrence of complications. The patient will be ready for surgery when the score ≥14 point. At this point the onset will be determined and so the patient can be transferred to the operating room .

If the patient experienced anxiety, propofol infusion (80-250 ug/kg/min) can be started. If the patient experienced pain during surgery the block considered failed and induction of general anesthesia should be started.

After end of the surgery the second investigator will continue to assess the patient for post operative pain every one hour for 24 hours to determine duration of the block.

DETAILED DESCRIPTION:
The purpose of this study to compare between three techniques( single- injection, intra-cluster -injection and double-injection) ultrasound-guided supraclavicular block of brachial plexus for surgery of forearm regarding onset of the block , duration, time of performance and possible complications

Study population & Sample size : 36 patients undergoing elective forearm surgeries in Kasr AL Aini Hospital will be included in the study , patients will be allocated in three groups 12 patient each.

Study Design : randomized comparative study , randomization will be done through closed opaque envelope

Methods :This study will be conducted at kasr al ainy Hospital Cairo university After obtaining ethics committee approval and written informed consent 36 patients (who will undergo surgery for forearm)included in the study classified into three groups Gs single injection technique ,Gic intra- cluster injection technique, Gd double injection technique For the 3 techniques , the investigator will prepare 20 gauge 10cm block needle and portable ultrasound machine (Siemens ACUSON X300 Ultrasound System with linear probe 8-14 MHZ).

In the preparation room, Standard monitors will be connected ,IV peripheral cannula will be inserted in upper limb contra lateral to surgical site and sedative e.g. midazolam 0.02mg/kg will be given. Patient will be positioned semi-sitting, the transducer is positioned in the transverse plane immediately superior to the clavicle at approximately its midpoint. Using a 3-cm, 27-gauge needle, 2 mL of local anesthetic is injected into the skin 1 cm lateral. In single-injection technique using in plane method and lateral to medial direction, local anesthetic (30 ml bupivacaine) is injected at the point where the subclavian artery meets the first rib. In intra- cluster-injection technique using in plane method and lateral to medial direction , the local anesthetic(30 ml bupivacaine) is injected inside main and satellite neural cluster.( Circumferential administration of local anesthetic rather than creating a single point injection ).

In double-injection technique using in plane method and lateral to medial direction half the volume of local anesthetic(15 ml bupivacaine) is injected at intersection of first rib and subclavian artery and another half(15 ml bupivacaine) is injected supero- lateral to subclavian artery to assure spread of the local anesthetic solution in all planes containing brachial plexus. the performance time will be recorded.

After block will be done, second investigator will examine the patient for sensory and motor block (every 10 minutes for 30 minutes) and for occurrence of complications. The patient will be ready for surgery when the score ≥14 point. At this point the onset will be determined and so the patient can be transferred to the operating room .

If the patient experienced anxiety, propofol infusion (80-250 ug/kg/min) can be started. If the patient experienced pain during surgery the block considered failed and induction of general anesthesia should be started.

After end of the surgery the second investigator will continue to assess the patient for post operative pain every one hour for 24 hours to determine duration of the block.

Possible Risks to study population : 1. Intravascular injection of local anaesthetic (if tip of needle is seen under ultrasound screen and the investigator is injecting local anaesthetic but nothing seen under ultrasound screen(tellet sign)) 2. Pneumothorax (asses pleura of the same side by chest x-ray after 6 hours) 3. Intraneural injection (keep an image or video of technique and seek for another opnion) Various studies demonstrated that if intraneural puncture occured the needle usually took a path away from the fascicles (intraneural perifascicular), while intraneural transfascicular puncture seemed relatively rare and intraneural intrafascicular placement of the needle even more uncommon. As long as the needle is placed intraneurally but in an extrafascicular fashion a safe injection and the absence of neurologic damage can be assumed.

4. Horner's syndrome (ptosis ,miosis ,anhydrosis may be due to involvement of cervical sympathetic plexus)

ELIGIBILITY:
Inclusion Criteria:

1. Age ( 18 -60 years)
2. ASA l & ASA II
3. Body mass index(20-35 Kg/m2)

Exclusion Criteria:

1. Pre-existing neuropathy
2. ASA lll & ASA lV
3. Previous operation in supraclavicular fossa
4. Coagulopathy
5. Allergy to local anesthetic
6. Pregnancy
7. Inability to visualize the brachial plexus during ultrasound scanning.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
onset of the block onset of anesthesia ( time in minutes from introduction of needle to appearance of 14 point score for motor and sensory block ) onset of the block | from 0- 25 minutes after complete injectio
  time in minutes from introduction of needle to appearance of 14 point score for motor and sensory block )

SECONDARY OUTCOMES:
Duration of the block | 25 minutes after injection till 6 hours post oprative
  from onset to appearance of pain in surgery site

OTHER OUTCOMES:
Complications | from injection till 24 hours postoprative
  intravascular injection , pneumothorax or horner syndrome
Time of first postoperative rescue analgesic | from injection till 24 hours postoprative
  the first time the patient ask for analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine CAIRO UNIVERISTY, Cairo, Egypt